CLINICAL TRIAL: NCT03694821
Title: Efficacy and Cost-effectiveness of Intra-Articular Ketorolac Injection for Knee Osteoarthritis: A Randomized, Controlled, Double-Blinded Study
Brief Title: Knee Injection RCT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: UConn Health (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-093-1
Record Dates: First submitted 2018-08-16; First posted 2018-10-03 (Actual); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee; Injection; Ketorolac
MeSH Terms: conditions — Osteoarthritis | interventions — Ketorolac Tromethamine; Methylprednisolone Acetate; hylan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ketorolac (Experimental): One knee injection of 2cc of ketorolac tromethamine (15mg/cc) in 5cc of 0.5% ropivacaine hydrochloride without epinephrine
  Interventions: Drug: Ketorolac Tromethamine Injection
- Corticosteroid (Active Comparator): One knee injection of 2 cc of methylprednisolone acetate (40mg/cc) in 5cc of 0.5% ropivacaine hydrochloride without epinephrine
  Interventions: Drug: Methylprednisolone Acetate Injection
- Hyaluronic Acid (Active Comparator): One knee injection of Hylan G-F 20 (Synvisc-One)
  Interventions: Drug: Hylan G-F 20

INTERVENTIONS:
Drug: Ketorolac Tromethamine Injection — One knee injection of 2cc of ketorolac tromethamine (15mg/cc) in 5cc of 0.5% ropivacaine hydrochloride without epinephrine
  Other Names: Ketorolac Tromethamine; NDC 63323-162-02; J Code J1885
  Arms: Ketorolac
Drug: Methylprednisolone Acetate Injection — One knee injection of 2 cc of methylprednisolone acetate (40mg/cc) in 5cc of 0.5% ropivacaine hydrochloride without epinephrine
  Other Names: DEPO-MEDROL; NDC 0009-3073-01; J Code J1030
  Arms: Corticosteroid
Drug: Hylan G-F 20 — One knee injection of Hylan G-F 20 (Synvisc-One)
  Other Names: Synvisc-One; NDC 58468-0090-03; J Code J7325
  Arms: Hyaluronic Acid

SUMMARY:
Hypothesis: Ketorolac injection is a cost-effective adjunct in the nonoperative treatment of knee osteoarthritis (OA) compared to steroids and viscosupplementation.

Aims/objectives: The objective of this randomized, controlled, double-blinded, prospective study is to assess the efficacy and cost-effectiveness of knee injection with ketorolac in the nonsurgical management of symptomatic OA compared to injections with corticosteroids and viscosupplements.

DETAILED DESCRIPTION:
The purpose of this research study is to examine the effectiveness of intra-articular (inside the joint) ketorolac injection compared to injection with either corticosteroid or hyaluronic acid for the treatment of painful knee osteoarthritis. Patients will be randomly assigned to receive either ketorolac (a nonsteroidal anti-inflammatory drug, methylprednisolone (a steroid), hyaluronic acid (a substance that is naturally present in the human body).

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who present with 1) symptomatic knee OA and radiographic evidence of joint space narrowing and 2) are interested in knee injections for pain relief.

Exclusion Criteria:

* Prior injections into the same knee within the past 6 months,
* Pregnant and/or lactating women,
* Inflammatory joint disease including rheumatoid or psoriatic arthritis,
* Concurrent use of anti-rheumatic drugs,
* Allergy or hypersensitivity to the study medications,
* Patients on an active pain management contract,
* Patients with insurance that requires pre-certification for any of the study drugs,
* Inability to make own decisions regarding the informed consent,
* Inability to read and/or understand English,
* Patients who are unable to return for follow-up or be reached by phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad J. Halawi, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dieppe PA, Lohmander LS. Pathogenesis and management of pain in osteoarthritis. Lancet. 2005 Mar 12-18;365(9463):965-73. doi: 10.1016/S0140-6736(05)71086-2. PMID 15766999
- [Background] Hootman JM, Helmick CG. Projections of US prevalence of arthritis and associated activity limitations. Arthritis Rheum. 2006 Jan;54(1):226-9. doi: 10.1002/art.21562. PMID 16385518
- [Background] Bone and Joint Initiative: The Burden of Musculoskeletal Diseases in the United States. http://www.boneandjointburden.org/2014-report/ivh12/osteoarthritis-and-allied-disorders
- [Background] Jevsevar DS. Treatment of osteoarthritis of the knee: evidence-based guideline, 2nd edition. J Am Acad Orthop Surg. 2013 Sep;21(9):571-6. doi: 10.5435/JAAOS-21-09-571. PMID 23996988
- [Background] Gray RG, Gottlieb NL. Intra-articular corticosteroids. An updated assessment. Clin Orthop Relat Res. 1983 Jul-Aug;(177):235-63. PMID 6345042
- [Background] Hunter DJ. Viscosupplementation for osteoarthritis of the knee. N Engl J Med. 2015 Mar 12;372(11):1040-7. doi: 10.1056/NEJMct1215534. No abstract available. PMID 25760356
- [Background] van der Weegen W, Wullems JA, Bos E, Noten H, van Drumpt RA. No difference between intra-articular injection of hyaluronic acid and placebo for mild to moderate knee osteoarthritis: a randomized, controlled, double-blind trial. J Arthroplasty. 2015 May;30(5):754-7. doi: 10.1016/j.arth.2014.12.012. Epub 2014 Dec 13. PMID 25548079
- [Background] Campbell KA, Erickson BJ, Saltzman BM, Mascarenhas R, Bach BR Jr, Cole BJ, Verma NN. Is Local Viscosupplementation Injection Clinically Superior to Other Therapies in the Treatment of Osteoarthritis of the Knee: A Systematic Review of Overlapping Meta-analyses. Arthroscopy. 2015 Oct;31(10):2036-45.e14. doi: 10.1016/j.arthro.2015.03.030. Epub 2015 May 19. PMID 25998016
- [Background] Berenbaum F. Osteoarthritis as an inflammatory disease (osteoarthritis is not osteoarthrosis!). Osteoarthritis Cartilage. 2013 Jan;21(1):16-21. doi: 10.1016/j.joca.2012.11.012. Epub 2012 Nov 27. PMID 23194896
- [Background] Brown GA. AAOS clinical practice guideline: treatment of osteoarthritis of the knee: evidence-based guideline, 2nd edition. J Am Acad Orthop Surg. 2013 Sep;21(9):577-9. doi: 10.5435/JAAOS-21-09-577. No abstract available. PMID 23996989
- [Background] Reuben SS, Connelly NR. Postoperative analgesia for outpatient arthroscopic knee sugery with intraarticular bupivacaine and ketorolac. Anesth Analg. 1995 Jun;80(6):1154-7. doi: 10.1097/00000539-199506000-00015. PMID 7762844
- [Background] Desai A, Ramankutty S, Board T, Raut V. Does intraarticular steroid infiltration increase the rate of infection in subsequent total knee replacements? Knee. 2009 Aug;16(4):262-4. doi: 10.1016/j.knee.2008.12.002. Epub 2009 Jan 12. PMID 19138855
- [Background] Jones AC, Pattrick M, Doherty S, Doherty M. Intra-articular hyaluronic acid compared to intra-articular triamcinolone hexacetonide in inflammatory knee osteoarthritis. Osteoarthritis Cartilage. 1995 Dec;3(4):269-73. doi: 10.1016/s1063-4584(05)80018-4. PMID 8689462
- [Background] Leardini G, Mattara L, Franceschini M, Perbellini A. Intra-articular treatment of knee osteoarthritis. A comparative study between hyaluronic acid and 6-methyl prednisolone acetate. Clin Exp Rheumatol. 1991 Jul-Aug;9(4):375-81. PMID 1934686
- [Background] Bellamy JL, Goff BJ, Sayeed SA. Economic Impact of Ketorolac vs Corticosteroid Intra-Articular Knee Injections for Osteoarthritis: A Randomized, Double-Blind, Prospective Study. J Arthroplasty. 2016 Sep;31(9 Suppl):293-7. doi: 10.1016/j.arth.2016.05.015. Epub 2016 May 18. PMID 27402605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Started | 4 | 8 | 6
Completed | 0 | 0 | 2
Not Completed | 4 | 8 | 4
Not completed — Study terminated | 4 | 8 | 4

BASELINE CHARACTERISTICS:
Population: Only age, sex, race and ethnicity data available. No other analysis completed due to study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid | Total
Number analyzed (Participants) | 4 | 8 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 4 | 14
  >=65 years | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 11
  Male | 2 | 3 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 3 | 7 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 4
  White | 3 | 4 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Pain Scale (VAS)
Description: average knee pain between 0 (no pain) and 10 (worst pain) 3 months following injection
Time Frame: 3 months post injection
Population: Data were collected, but the PI has left the institution. All efforts to locate and analyze the data have been exhausted; therefore no data are available to report.
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: self-reported pain, stiffness and functioning
Time Frame: 3 and 6 months post injection
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Oxford Knee Questionnaire
Description: self-reported pain, stiffness and functioning
Time Frame: 3 and 6 months post injection
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Koos, Jr. Knee Survey
Description: self-reported pain, stiffness and functioning
Time Frame: 3 and 6 months post injection
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Visual Analogue Pain Scale (VAS)
Description: average knee pain between 0 (no pain) and 10 (worst pain) 6 months following injection
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Patient Satisfaction
Description: satisfaction with treatment rated as "Yes" or "No"
Time Frame: 3 and 6 months post injection
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Non-routine Visits Due to Inadequate Pain Relief or Complications
Description: Any additional visits due to inadequate pain relief or complications
Time Frame: 3 months post injection
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Cost of Intervention
Description: cost of each injection
Time Frame: 3 months post injection
Population: as for outcome 1
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: Same definition was used.
Arm/Group | Ketorolac | Corticosteroid | Hyaluronic Acid
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 1/4 | 0/8 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac (N=4) | Corticosteroid (N=8) | Hyaluronic Acid (N=6)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03694821/Prot_SAP_000.pdf